CLINICAL TRIAL: NCT06051643
Title: Use of Motor Rehabilitation Courses in Children With Cerebral Palsy in 2022
Brief Title: Use of Motor Rehabilitation Courses in Children With Cerebral Palsy
Acronym: ERSRMPC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0023
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Children; Motor rehabilitation course; Survey and Questionnaire
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2022, the prevalence of Cerebral Palsy (CP) is 2.5 cases per 1000 live births. In France, 125,000 persons are affected by CP. Many treatments and therapies exist to reduce CP-related disorders, but CP remains uncurable. Motor Rehabilitation Courses (MRC) are one of those therapies used with children with CP. Their uses has not been studied in France yet.

The aim of this survey is to find out about the use of motor rehabilitation courses for children with CP and, where appropriate, the content of these courses. This questionnaire will be used to determine the use and different types of MRS in which children participate.

DETAILED DESCRIPTION:
In total, the questionnaire contains 131 items divided into 13 groups. The estimated filling time is 20 minutes.

The questionnaire is divided as follows:

1. INFORMATION DOCUMENT FOR THE RESEARCH PARTICIPANT
2. About the person with cerebral palsy
3. About the respondent
4. About the usual motor rehabilitation
5. About participation in motor rehabilitation courses
6. 7) 8) Information about MRS

9) Relationship of care or treatment received to participation in MRS 10) Information about the child 11) Information about the child's environment 12) Additional comments from the respondent regarding the MRS 13) Respondent's opinion on the questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Child with a diagnosis of cerebral palsy
* Aged between 6 and 18 years

Exclusion Criteria:

* Child diagnosed with CP after age 6
* Between 1 and 6 years of age

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Represents children with cerebral palsy aged 6 to 18
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the use of motor rehabilitation courses in children with cerebral palsy | Each participant will answer for 20 minutes an expert-validated questionnaire on the internet once recruited in the study
  Prevalence of the use of motor rehabilitation courses